CLINICAL TRIAL: NCT00912288
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled 26-Week Trial To Evaluate The Efficacy And Safety Of Dimebon In Patients With Moderate-To-Severe Alzheimer's Disease
Brief Title: A Phase 3 Efficacy Study Of Dimebon In Patients With Moderate To Severe Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1451006
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease moderate-to-severe memantine safety and efficacy
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dimebon (Experimental)
  Interventions: Drug: Dimebon 20 mg po TID
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo po TID

INTERVENTIONS:
Drug: Dimebon 20 mg po TID — Dimebon 10 mg po TID for 1 week followed by Dimebon 20 mg TID for 25 weeks
  Other Names: PF-01913539; Latrepirdine Dihydrochloride
  Arms: Dimebon
Drug: Placebo po TID — Placebo (matched to Dimebon) po for 26 weeks
  Arms: Placebo

SUMMARY:
No Dimebon clinical data exist yet in patients with disease that has advanced to the moderate-to-severe stage. Therefore, this study evaluates the safety and efficacy of Dimebon in patients with moderate-to-severe AD who are receiving existing background therapy with memantine.

DETAILED DESCRIPTION:
This study was terminated on May 7, 2010 due to modification of the dimebon development plan following the lack of demonstration of efficacy in the completed DIM14 (CONNECTION) Study. The study was not terminated due to any safety findings. Dimebon has been well-tolerated in clinical trials. Demonstration of efficacy for dimebon in Alzheimer's disease is pending completion of the ongoing DIM18 (CONCERT) Study.

ELIGIBILITY:
Inclusion Criteria:

* Are men and women ≥ 50 years of age with a diagnosis of Alzheimers disease.
* Have a Mini-Mental State Exam between 5 and 14 inclusive.
* Have been taking the medication memantine (ie., Namenda) for at least six months prior to this study.
* Must have a caregiver who assists the patient at least five days per week for at least three hours per day, who can accompany patient to study visits, and who has an intimate knowledge of the patient's health states and personal care.

Exclusion Criteria:

* Have taken medicines for Alzheimers disease other than memantine (e.g., donepezil, rivastigmine, galantamine, tacrine) within 2 months prior to this study.
* Dementia other than Alzheimers disease.
* Any medical condition or reason that interferes with the ability of the patient to participate in or complete the trial or places the patient at undue risk, as judged by the study doctor.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (20):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Delray Beach, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Cordova, Tennessee
  - Pfizer Investigational Site, Middleton, Wisconsin
- Canada (3):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Günzburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Mittweida
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Székesfehérvár
- Portugal (2):
  - Pfizer Investigational Site, Amadora
  - Pfizer Investigational Site, Coimbra
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Michalovce
  - Pfizer Investigational Site, Rožňava
  - Pfizer Investigational Site, Žilina
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Algorta, Getxo, Bilbao
  - Pfizer Investigational Site, Salt, Girona
  - Pfizer Investigational Site, Seville, Sevilla
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Kocaeli
  - Pfizer Investigational Site, Samsun

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451006&StudyName=A%20Phase%203%20Efficacy%20Study%20Of%20Dimebon%20In%20Patients%20With%20Moderate%20To%20Severe%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimebon: Dimebon (latrepirdine) 10 milligram (mg) tablet orally three times a day for 1 week (titration period), followed by dimebon (latrepirdine) 20 mg tablet orally three times a day up to Week 26.
- Placebo: Placebo tablet matched to 10 mg of dimebon (latrepirdine) tablet orally three times a day for 1 week (titration period), followed by placebo tablet matched to 20 mg dimebon (latrepirdine) tablet orally three times a day up to Week 26.
Period: Overall Study
Arm/Group | Dimebon | Placebo
Started | 44 | 42
Completed | 3 | 2
Not Completed | 41 | 40
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Study terminated by sponsor | 34 | 35
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dimebon | Placebo | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Customized [Number; unit: Participants]
  50 to 59 years | 2 | 1 | 3
  60 to 69 years | 9 | 8 | 17
  70 to 79 years | 20 | 16 | 36
  80 to 85 years | 10 | 9 | 19
  Greater than 85 years | 3 | 8 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Severe Impairment Battery (SIB) Score at Week 26
Description: SIB developed for evaluation of cognitive function in participants, who demented to a degree that they cannot complete conventional neuropsychological testing. Test items consisted of simple, one-step commands presented with gestural cues and instructions that were repeated if necessary. SIB test consisted of 51-item scale, divided into 9 subscales: social interaction (0-6), memory (0-14), orientation (0-6), language (0-46), attention (0-6), praxis(0-8), visuospatial ability(0-8), construction(0-4), orienting to name(0-2). Total possible score:0-100; lower score = greater cognitive impairment.
Time Frame: Baseline, Week 26
Population: Data for this outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis due to early termination of the study.
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (Severe) (ADCS-ADLsev) Score at Week 26
Description: ADCS-ADLsev: 19-item scale measures basic and instrumental abilities in participant population and had good metric properties and reliability in detecting change. Individual score range: 0 to 5 for telephone, 0 to 4 for dressing, watch television, get around outside home, 0 to 3 for eating, walking, toilet, bathing, grooming, conversation/small talk, clear dishes, find personal belongings, obtain beverages, dispose of garbage, left on own, 0 to 1 for run water from and turn off faucet to wash hands, turn on and off light. Total score range: 0 to 54 lower scores=greater functional impairment.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in the Neuropsychiatric Inventory (NPI) Total Score at Week 26
Description: NPI:12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, nighttime behavior. Severity(1=Mild to 3=Severe),frequency(1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score(range 0-12). Total score=sum of each domain score(range 0-144);higher score=greater behavioral disturbances;negative change score from baseline=improvement.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Sum of the Delusions and Hallucinations Sub-domain Scores of the NPI
Description: NPI is a 12-domain caregiver assessment of behavioral disturbances occurring in dementia. Severity (1=Mild to 3=Severe) and frequency (1=occasionally to 4=very frequently) scales were recorded separately for each domain and their product gives individual domain score (range 0-12). Sum of delusions and hallucinations sub-domain scores of NPI was calculated as a measure of Alzheimer's Disease (AD) related psychosis. Total possible score range: 0-24 with higher score indicating greater behavioral disturbances.
Time Frame: Week 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in the Mini-Mental State Examination (MMSE) Score at Week 26
Description: MMSE measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. Total score derived from sub-scores; total ranged from 0 to 30, higher score indicates better cognitive state.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC-plus) Scores
Description: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) version of CIBIC-Plus was used to assess participant's overall disease severity. The corresponding baseline assessment rated participant on 7-point scale: (1) extremely severe AD to (7) no symptoms of AD. Overall impression of change from baseline was rated on a 7-point scale: 1=marked improvement; 2=moderate improvement; 3=minimal improvement; 4=no change; 5=minimal worsening; 6=moderate worsening; 7=marked worsening; all assessments are relative to baseline. Higher score = worsening of global function.
Time Frame: Week 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Resource Utilization in Dementia-Lite Version (RUD-Lite)
Description: RUD Lite: instrument used to assess amount of both formal and informal resources used by demented participants and primary caregiver. It was completed by caregivers and compiles data on following resources: use of social services, frequency and duration of hospitalizations, all contacts with health care professionals, participant living accommodations, amount of time the caregiver spends giving care and the impact of care giving on the caregiver's job. Overall cost of care was evaluated to quantify resources utilized.
Time Frame: Baseline, Weeks 12, 18, 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Euro Quality of Life - 5 Domain (EQ-5D) Assessment
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Total possible score ranged from 5 to 15; lower score indicated a better health state.
Time Frame: Baseline, Weeks 12, 26
Population: as for outcome 1
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Population Pharmacokinetic (PK) Analysis
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Pre-dose, 0.5 to 1.5 hours, 2.5 to 3.5 hours post-dose at Week 12
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Any untoward medical occurrence (including clinially important changes in clinical safety laboratory assessments, electrocardiograms and vital signs) in a participant who received study treatment was considered an AE without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 30 (follow-up)
Population: Safety analysis set included all participants who received at least 1 dose of study medication, including partial doses.
Measure: Number; unit: Participants
Arm/Group | Dimebon | Placebo
Number analyzed (Participants) | 44 | 42
Participants | 27 | 18

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dimebon | Placebo
Serious Adverse Events (participants affected / at risk) | 4/44 | 3/42
Other Adverse Events (participants affected / at risk) | 10/44 | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=44) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dimebon (N=44) | Placebo (N=42)
Nausea (Gastrointestinal disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 3
Urinary tract infection (Infections and infestations) | 5 | 2
Agitation (Psychiatric disorders) | 5 | 2

LIMITATIONS AND CAVEATS:
Results are not summarized because of early termination of the study due to modification in the development plan of the study medication following lack of demonstration of efficacy in the completed DIM14 CONNECTION (B1451002/NCT00675623) study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.